CLINICAL TRIAL: NCT04641858
Title: BCG Vaccine to Reduce Unplanned Absenteeism Due to Illness of Health Care Workers During the COVID-19 Pandemic. A Multi-center Randomised Controlled Trial (BCG-COVID-RCT)
Brief Title: BCG to Reduce Absenteeism Among Health Care Workers During the COVID-19 Pandemic
Acronym: EDCTP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Institute of Hygiene and Tropical Medicine, NOVA University, Lisbon, Portugal (Unknown); University of Cape Verde, Praia, Cape Verde (Unknown); National Institute of Public Health of Cape Verde, Praia, Cape Verde (Unknown); Centro de Investigacao em Saude de Manhica (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Bandim Health Project, Bissau, Guinea-Bissau (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCG-COVID-RCT
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Covid19; Morbidity; Absenteeism
Keywords: Innate immune training; Non-specific effects of BCG; Heterologous effects
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multi-center randomized placebo-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to treatment. The physicians administering the BCG vaccine or placebo will not be blinded. Those assessing outcomes will be blinded to the randomization allocation. In case of serious adverse events, the participant can be unblinded after consultation with the coordinating PI or sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG-Denmark (Active Comparator): Participants that are randomized in the active arm will receive an adult 0.1 ml dose of BCG vaccine (BCG-Denmark, AJ Vaccines) in the skin covering the right upper deltoid muscle. Each 0.1 ml vaccine contains between 200000 to 800000 colony forming units of the live attenuated strain of Mycobacterium bovis (BCG), Danish strain 1331.
  Interventions: Biological: BCG-Denmark
- Control (Placebo Comparator): Placebo will be 0.1 ml sterile 0.9 % NaCl, which has a similar color and appearance as the resuspended BCG vaccine.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: BCG-Denmark — Participants randomized to receive BCG will receive one 0.1 ml dose of Mycobacterium bovis BCG live attenuated BCG-Denmark vaccine (AJ Vaccines, Copenhagen, Denmark) by intradermal injection in the left deltoid region.
  Arms: BCG-Denmark
Biological: Saline — Participants randomized to the control group will receive one 0.1 ml dose sterile 0.9 % NaCl by intradermal injection in the right deltoid region.
  Arms: Control

SUMMARY:
The COVID-19 pandemic challenges available hospital capacity. Strategies to protect health care workers (HCW) are desperately needed. Bacille Calmette- Guérin (BCG) has protective non-specific effects against other infections; a plausible immunological mechanism has been identified in terms of "trained innate immunity".

The primary objective of the study is to evaluate whether BCG can reduce unplanned absenteeism due to illness among HCW during the COVID-19 pandemic. Secondary objectives are to reduce the number of HCW that are infected with COVID-19, reduce hospital admissions for HCW and to improve the capacity for clinical research.

Design: Single-blind, parallel-group placebo-controlled multi-centre block randomized trial including a total of 1050 HCW. The study sites will be the Manhiça hospital in Mozambique, Central Hospital Dr. Agostinho Neto and Central Hospital Dr. Baptista de Sousa in Cape Verde and Hospital Nacional Simão Mendes and other hospitals in the capital Bissau in Guinea-Bissau. Population: HCW (nurses/physicians/others) ≥18 years.

Intervention: Block randomization 1:1 to intradermal standard dose (0.1 ml) of BCG vaccine or placebo (saline). Endpoints: Primary: Days of unplanned absenteeism due to illness. Secondary: Days of absenteeism because of documented COVID-19; cumulative incidence of infectious disease hospitalizations.

Follow-up: mobile phone interviews every second week, regarding symptoms, absenteeism and causes, COVID-19 testing (if done) and their results.

Perspectives: If BCG can reduce HCW absenteeism it has global implications. The intervention can quickly be scaled up all over the world.

DETAILED DESCRIPTION:
The main hypothesis for this study is that BCG vaccination of HCW reduces unplanned absenteeism due to illness by 20%.

Trial design Single-blind, parallel-group placebo-controlled adaptive multicentre trial, with block-randomisation 1:1 (treatment:placebo) in blocks of 20 within strata defined by gender (male/female) and occupational group (doctors/ nurses/other) to an intradermal standard 0.1 ml dose of BCG vaccine or placebo (saline) including a total of 1050 HCW (BCG arm and placebo arm).

Study population:

Health Care Workers defined as a person who delivers care and services to the sick and ailing either directly as doctors and nurses or indirectly as aides, helpers, laboratory technicians, or even medical waste handlers.

Intervention:

The intervention will consist of the administration of an intradermal injection of a standard 0.1 ml adult dose of attenuated Mycobacterium bovis BCG (Bacillus Calmette-Guerin), Danish strain 1331, 2-8 × 10*5 CFU or the placebo comparator: intradermal standard 0.1 ml saline solution (NaCl 0.9%). Both BCG and saline solution will be injected in the skin over the upper deltoid muscle.

Blinding:

The BCG vaccine will be administered by study physicians/nurses, who are not blinded but also not involved in the data collection. Participants, data collectors and data entry clerks will be blinded to the treatment allocation.

In case of serious adverse events, the participant can be unblinded after consultation with the investigator or the vaccinating physician/nurse. When the study has ended, all participants will receive information about the intervention that they received.

Follow-up:

Follow-up will last for 6 months (182 days). Every second week, participants will be contacted over telephone and interviewed for symptoms and absenteeism from work. By the end of follow-up, participants will be invited for another POC test for COVID-19 serology.

Sample size:

The sample size was calculated on the basis of the primary hypothesis. A total of 1050 HCW randomized with an estimated loss to follow-up of 5%, and a mean number of days off work due to illness in the control group of 5 days (SD=5) over a 6-month period will demonstrate a reduction among BCG vaccinated of 20% for a mean absence of 4 days (80% power and alpha 0.05). The estimated loss to follow-up (5%) was based on past telephone-based surveys conducted in Mozambique and Bissau.

ELIGIBILITY:
Inclusion Criteria:

* health care worker (physician, nurse, or other) based at one of the research hospitals.
* age ≥18 years

Exclusion Criteria:

* known allergy to (components of) BCG or serious adverse events to prior BCG administration;
* known previous, active or latent infection with Mycobacterium tuberculosis or other mycobacterial species
* fever (>38 C) within past 24 hours;
* previous confirmed COVID-19 (positive test - PCR or antibody);
* suspicion of active viral or bacterial infection
* severely immunocompromised subjects
* self-reported HIV infection
* self-reported pregnancy;
* active solid or non-solid malignancy or lymphoma within the prior two years;
* contraindications for live attenuated vaccine administration.
* not having a mobile phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Days of unplanned absenteeism due to illness | 6 months after inclusion
  Unplanned absenteeism is defined by being absent from work due to causes other than holidays, parental leave, and other planned leaves, family assistance (including mourning leave) and quarantine measures.

SECONDARY OUTCOMES:
Days of unplanned absenteeism due to documented COVID-19 | 6 months after inclusion
  Unplanned absenteeism is defined by being absent from work due to causes other than holidays, parental leave, and other planned leaves, family assistance (including mourning leave) and quarantine measures.
Cumulative incidence of hospital admissions due to illness (minus accidents). | 6 months after inclusion
  Hospital admissions involves staying at a hospital for at least one night or more for medical reasons. It includes admissions to hospital wards and overnight stays in emergency departments.
Death | 6 months after inclusion
  Whether the participant died during follow-up

OTHER OUTCOMES:
Hospitalisation for COVID-19 | 6 months after inclusion
  Refers to the number of nights of hospitalisation due to COVID-19
Hospitalisation besides COVID-19 | 6 months after inclusion
  Refers to the number of nights of hospitalisation due to other reasons besides COVID-19
Time to hospitalisation | 6 months after inclusion
  Time, in days, from enrolment to first night of hospitalisation
Time to absenteeism | 6 months after inclusion
  Time, in days, from enrolment to first day absent from work due to ill-health and disease
Time to COVID-19 absenteeism | 6 months after inclusion
  Refers to the number of days since enrolment to first day absent from work due to suspected COVID-19
COVID-19 infection | 6 months after inclusion
  Describes if the participant is positive for SARS-CoV2 or has had COVID-19
Time to COVID-19 | 6 months after inclusion
  Time, in days, from enrolment to positive test for SARS-CoV2

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stabell Benn, Professor, Principal Investigator — University of Southern Denmark
Locations (2):
- Bandim Health Project, Bissau, SAB, Guinea-Bissau
- Manhiça Health Research Centre, Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual data can be shared on the basis of a data sharing proposal sent to professor Inês Fronteira ifronteira@ihmt.unl.pt
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When follow-up has been completed and the dataset have been closed.
Access Criteria: Non-identifiable individual data can be shared on the basis of a data sharing proposal sent to ifronteira@ihmt.unl.pt

REFERENCES:
- [Background] Aaby P, Kollmann TR, Benn CS. Nonspecific effects of neonatal and infant vaccination: public-health, immunological and conceptual challenges. Nat Immunol. 2014 Oct;15(10):895-9. doi: 10.1038/ni.2961. PMID 25232810
- [Background] Aaby P, Benn CS. Developing the concept of beneficial non-specific effect of live vaccines with epidemiological studies. Clin Microbiol Infect. 2019 Dec;25(12):1459-1467. doi: 10.1016/j.cmi.2019.08.011. Epub 2019 Aug 23. PMID 31449870
- [Background] Benn CS, Fisker AB, Rieckmann A, Sorup S, Aaby P. Vaccinology: time to change the paradigm? Lancet Infect Dis. 2020 Oct;20(10):e274-e283. doi: 10.1016/S1473-3099(19)30742-X. Epub 2020 Jul 6. PMID 32645296
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Rieckmann A, Villumsen M, Sorup S, Haugaard LK, Ravn H, Roth A, Baker JL, Benn CS, Aaby P. Vaccinations against smallpox and tuberculosis are associated with better long-term survival: a Danish case-cohort study 1971-2010. Int J Epidemiol. 2017 Apr 1;46(2):695-705. doi: 10.1093/ije/dyw120. PMID 27380797
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Benn CS, Fisker AB, Whittle HC, Aaby P. Revaccination with Live Attenuated Vaccines Confer Additional Beneficial Nonspecific Effects on Overall Survival: A Review. EBioMedicine. 2016 Aug;10:312-7. doi: 10.1016/j.ebiom.2016.07.016. Epub 2016 Jul 15. PMID 27498365
- [Background] Roth AE, Benn CS, Ravn H, Rodrigues A, Lisse IM, Yazdanbakhsh M, Whittle H, Aaby P. Effect of revaccination with BCG in early childhood on mortality: randomised trial in Guinea-Bissau. BMJ. 2010 Mar 15;340:c671. doi: 10.1136/bmj.c671. PMID 20231251
- [Background] Biot C, Rentsch CA, Gsponer JR, Birkhauser FD, Jusforgues-Saklani H, Lemaitre F, Auriau C, Bachmann A, Bousso P, Demangel C, Peduto L, Thalmann GN, Albert ML. Preexisting BCG-specific T cells improve intravesical immunotherapy for bladder cancer. Sci Transl Med. 2012 Jun 6;4(137):137ra72. doi: 10.1126/scitranslmed.3003586. PMID 22674550
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT04641858/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT04641858/SAP_001.pdf